CLINICAL TRIAL: NCT02124863
Title: Influence of Intrapulmonary Percussive Ventilation (IPV) on Gastro-oesophageal Reflux (GOR) in Infants From 0 to 12 Months.
Brief Title: Influence of IPV on GOR in Infants From 0 to 12 Months.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Filip Van Ginderdeuren, PT, Drs, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVG002
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Gastro-oesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intrapulmonary Percussive Ventilation (Experimental): number of refluxes during 20 min of IPV ( rate : 300/min, p = 10cmH2O) at least 120 min after feeding
  Interventions: Device: Intrapulmonary Percussive Ventilation

INTERVENTIONS:
Device: Intrapulmonary Percussive Ventilation — 20 min IPV freq 300/min, p 10cmH2O

SUMMARY:
The purpose of this study is to determine whether Intrapulmonary Percussive Ventilation ( airway clearance technique) provokes or aggravates gastro-oesophageal reflux in infants from 0 to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* infants from 0 to 12 months
* impedance monitoring

Exclusion Criteria:

* gestational age < 24w
* anti-reflux medication
* Nissen fundoplication
* no parental consent

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: fili van ginderdeuren, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intrapulmonary Percussive Ventilation
Started | 67
Completed | 50
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | Intrapulmonary Percussive Ventilation
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50
  Between 18 and 65 years | 0
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 25
  Male | 25
Region of Enrollment [Number; unit: participants]
  Belgium | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Refluxes
Description: Every two hours after feeding, the number of refluxes during 20 minutes are measured. The mean number of refluxes during these periods were calculated and compared to the number of refluxes during 20 minutes of IPV
Time Frame: during 20 minutes of IPV compared to mean number of refluxes during 20 minutes.
Population: All patients receiving IPV were their own controls
Measure: Mean (Standard Deviation); unit: number of refluxes
Groups:
- Control: mean number of refluxes during 20 min, 120 min after each meal
Arm/Group | Intrapulmonary Percussive Ventilation | Control
Number analyzed (Participants) | 50 | 50
number of refluxes | 0.48 (0.76) | 0.97 (0.95)

ADVERSE EVENTS:
Time Frame: 20 minutes
Description: during treatment
Arm/Group | Intrapulmonary Percussive Ventilation | Control
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67
Other Adverse Events (participants affected / at risk) | 0/67 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No